CLINICAL TRIAL: NCT01326000
Title: A Randomized, Multicenter, Open-label Phase II Study of RO5083945 in Combination With FOLFIRI Versus FOLFIRI Plus Cetuximab or FOLFIRI Alone as Second Line Treatment in Patients With KRAS Wild-type or Mutant Metastatic Colorectal Cancer
Brief Title: A Study of RO5083945 in Combination With FOLFIRI Versus FOLFIRI Plus Cetuximab or FOLFIRI Alone as Second Line Treatment in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP25438
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol; imgatuzumab; Cetuximab

ARMS (4):
- KRAS WT A (Experimental)
  Interventions: Drug: FOLFIRI; Drug: RO5083945
- KRAS WT B (Active Comparator)
  Interventions: Drug: FOLFIRI; Drug: cetuximab
- KRAS mutant A (Experimental)
  Interventions: Drug: FOLFIRI; Drug: RO5083945
- KRAS mutant B (Active Comparator)
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: FOLFIRI — standard iv chemotherapy
Drug: RO5083945 — 1400 mg iv on Day 1 and Day 8, and every 2 weeks thereafter
  Arms: KRAS WT A; KRAS mutant A
Drug: cetuximab — 400 mg/m2 iv on Day 1, followed by 250 mg/m2 iv every week
  Arms: KRAS WT B

SUMMARY:
This randomized, multicenter, open label study will evaluate the safety and efficacy of RO5083945 in combination with FOLFIRI as compared to FOLFIRI plus cetuximab or FOLFIRI alone as second line treatment in patients with metastatic colorectal cancer. Patients will be randomized to receive RO5083945 (1400 mg intravenously on Day 1 and Day 8 and every 2 weeks thereafter) plus FOLFIRI standard iv chemotherapy or FOLFIRI plus cetuximab (400 mg/m2 iv on Day 1 followed by 250 mg/m2 iv every week) or FOLFIRI alone. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Carcinoma of the colon and/or rectum
* Disease progression during or within 6 months of last dose of oxaliplatin containing first-line combination therapy for metastatic disease
* ECOG performance status 0-1
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Prior treatment with monoclonal antibody/small molecule against epidermal growth factor receptor (EGFR)
* Prior treatment with irinotecan
* Radiotherapy within the last 4 weeks before first dose of study drug (except for limited field palliative radiotherapy for bone pain relief)
* CNS metastasis
* History of or active autoimmune disorders/conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival: tumour assessments by CT scan or MRI according to RECIST criteria | approximately 18 months

SECONDARY OUTCOMES:
Overall Response Rate: tumour assessments by CT scan or MRI according to RECIST criteria | approximately 18 months
Duration of response: time from complete or partial response to disease progression or death | approximately 18 months
Clinical benefit rate: stable disease for >6 weeks, complete response or partial response; tumour assessments by CT scan or MRI according to RECIST criteria | approximately 18 months
Overall survival | approximately 18 months
Safety: Incidence of adverse events | approximately 18 months
Effect of concomitant FOLFIRI on pharmacokinetics of RO5083945 and vice versa | approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- United States (14):
  - Encinitas, California
  - Highland, California
  - La Jolla, California
  - La Verne, California
  - Los Angeles, California
  - San Diego, California
  - Harvey, Illinois
  - Skokie, Illinois
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Sayre, Pennsylvania
  - Greenville, South Carolina
  - Memphis, Tennessee
- Australia (6):
  - Newcastle, New South Wales
  - Port Macquarie, New South Wales
  - Adelaide, South Australia
  - Box Hill, Victoria
  - EAST Bentleigh, Victoria
  - Frankston, Victoria
- Belgium (4):
  - Brussels
  - Edegem
  - Ghent
  - Leuven
- France (6):
  - Bordeaux
  - Brest
  - Lille
  - Paris
  - Saint-Herblain
  - Toulouse
- Germany (6):
  - Essen
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Regensburg
- Italy (5):
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Milan, Lombardy
  - Pavia, Lombardy
- Poland (2):
  - Olsztyn
  - Szczecin
- Spain (6):
  - Sabadell, Barcelona, Barcelona
  - Santander, Cantabria
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- United Kingdom (10):
  - Aberdeen
  - Belfast
  - Bournemouth
  - Cardiff
  - Dorchester
  - Glasgow
  - London
  - Northwood
  - Romford
  - Weston-super-Mare